CLINICAL TRIAL: NCT00313755
Title: Back-to Back Trial of Narrow Band Imaging (NBI) With Magnification Versus Standard Colonoscopy for Colonic Neoplasia Surveillance in Hereditary Non-Polyposis Colorectal Cancer (HNPCC) Patients
Brief Title: Magnification Narrow Band Imaging Colonoscopy for Hereditary Non-Polyposis Colorectal Cancer Surveillance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 06/NBI5/15
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2006-11

CONDITIONS: Colorectal Neoplasms, Hereditary Nonpolyposis
Keywords: colonoscopy, narrow band imaging,; high definition endoscopy; colorectal cancer; dysplasia; hereditary non-polyposis colorectal cancer; Lynch Syndrome; HNPCC
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms | interventions — Narrow Band Imaging

INTERVENTIONS:
Procedure: Narrow Band Imaging

SUMMARY:
The purpose of this study is to determine whether a new colonoscopic viewing technique called narrow band imaging (NBI)can help doctors detect more patients with at least one pre-cancerous area than conventional colonoscopy using white light alone in patients with genetically inherited high risk for bowel cancer (HNPCC).

DETAILED DESCRIPTION:
Colorectal cancer is the second commonest cause of cancer death. Some people have an inherited defect in the genes which repair DNA which results in a very high risk of colorectal (bowel) cancer at a young age. This syndrome is called hereditary non-polyposis colorectal cancer (HNPCC) or Lynch syndrome. Colonoscopic surveillance of HNPCC patients has been shown to reduce the risk of colorectal cancer and allow detection at an earlier stage, but even with meticulous examination, some precancerous lesions or cancers are missed.

Precancerous lesions in HNPCC are difficult to see and may be advanced even if as small as a few millimeters. Endoscopists have used spraying dye on the lining of bowel (Chromoendoscopy) successfully to improve detection of abnormal areas; however this is time consuming and requires extra time and equipment and despite the benefits seen in two studies is not widely used in routine clinical practice in the UK.

Narrow Band Imaging (NBI) is a technique that relies on light to improve contrast for the smallest blood vessels in the bowel lining which shows up precancerous areas as they have a richer vascular network. It is sometimes described as "digital chromoendoscopy" as the images produced are similar to chromoendoscopy, but it is much simpler and quicker to use. With magnification it allows assessment of the fine mucosal surace pattern (pit pattern) of lesion which allows an assessment of their likelihood of being precancerous. Autofluorescence endoscopy uses short wavelength light and light filters to produce a false colour image of the bowel lining where polyps stand out. These techniques have been used with some success in the oesophagus and stomach but little work is available for the colon.

We aim to see if NBI with magnification is better than standard colonoscopy for detecting precancerous areas. This is likely as it produces images similar to chromoendoscopy which is already shown to help. If a potentially precancerous area is found we will use other types of endoscopy, in particular NBI and autofluorescence to see if these techniques are helpful for discriminating between pre-cancerous and non-cancerous areas.

ELIGIBILITY:
Inclusion Criteria:

* patients with HNPCC according to the Amsterdam II criteria
* patients over 18 years

Exclusion Criteria:

* pregnant patients
* unable or unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with at least one adenoma
after white light endoscopy compared with the number of patients
with at least one adenoma after white light NBI in the right colon.

SECONDARY OUTCOMES:
Total number of lesions detected with white light vs NBI.
Number of advanced neoplasm detected with white light vs NBI.
Number of hyperplastic polyps detected by white light vs NBI.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Saunders, MD FRCP, Study Director — London North West Healthcare NHS Trust
Locations (1):
- North West London Hospitals NHS Trust - St Mark's, London, Middlesex, United Kingdom

REFERENCES:
- [Derived] East JE, Suzuki N, Stavrinidis M, Guenther T, Thomas HJ, Saunders BP. Narrow band imaging for colonoscopic surveillance in hereditary non-polyposis colorectal cancer. Gut. 2008 Jan;57(1):65-70. doi: 10.1136/gut.2007.128926. Epub 2007 Aug 6. PMID 17682000